CLINICAL TRIAL: NCT00168610
Title: Should Infants Receive High-dose Vitamin A Supplementation With BCG Vaccine at Birth in Developing Countries? Randomized Prospective Studies in Guinea-Bissau
Brief Title: Vitamin A Supplementation With Bacille Calmette Guerin (BCG) Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Collaborators: March of Dimes (Other); Leiden University Medical Center (Other); Medical Research Council Unit, The Gambia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6-FY04-51-VITA2; 6-FY04-51
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Infant Mortality; Morbidity
Keywords: Vitamin A; BCG; Infant mortality; Morbidity; Low-income country; Mortality
MeSH Terms: conditions — Infant Death | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
In the present study the investigators wish to address the effects of different doses of vitamin A supplementation in low and normal birth weight infants.

Hypotheses:

* Vitamin A supplementation administered at birth together with BCG vaccination is associated with a 30% reduction in infant mortality and morbidity during the first year of life in both normal and low birth weight infants.
* A lower dose of vitamin A may be even more beneficial than a high dose.

DETAILED DESCRIPTION:
Vitamin A deficiency is common in low-income countries. Vitamin A supplementation to children above 6 months of age reduces all-cause mortality by 23% to 30%. Studies on vitamin A supplementation in infants younger than 6 months of age have reported inconsistent effects on mortality. Studies providing supplementation between 1 and 5 months of age have found no effect or even a negative effect. However, the only two studies of supplementation at birth, both conducted in Asia, showed substantial significant reductions in infant all-cause mortality.

The beneficial effect of neonatal vitamin A supplementation may be a result of correcting the congenital vitamin A deficiency resulting from maternal vitamin A deficiency. On the other hand, it has been speculated that the beneficial effect of vitamin A supplementation given at birth may in part be explained by a synergistic effect of vitamin A supplementation and BCG vaccination given at the time of birth.

The protective effect on mortality of vitamin A supplementation given at birth needs to be confirmed in an African population. Furthermore, none of the two previous studies have reported data on the vaccination status of the included infants.

In the proposed studies, the effect on mortality and morbidity of giving vitamin A supplementation simultaneously with BCG vaccination at birth to both normal and low birth weight infants will be investigated in an African population. Furthermore, the effects of vitamin A supplementation will be evaluated with respect to effect on growth, the response to BCG vaccination, infant vitamin A status and infant cytokine profile, malaria, measles, rotavirus infection and RSV infection. The mechanisms behind the effects of vitamin A will be evaluated. The potential interactions between vitamin A, sex and vaccines will be taken into account in all analyses.

This will be done in two studies of newborn children. Study A includes 6,000 normal birth weight infants (> 2500 g) randomized to 50,000 or 25,000 IU vitamin A or placebo given simultaneously with BCG vaccine. Study B includes 1,600 low birth weight infants (< 2500 g) randomized to vitamin A or placebo and early BCG or late BCG in a two-by-two factorial design. The studies take place in Guinea-Bissau, West Africa. The study area consists of five districts in the capital of Guinea-Bissau. The Bandim Health Project has been working in the study area for almost 25 years, and a demographic surveillance system has been established and has functioned for many years.

ELIGIBILITY:
Inclusion Criteria:

* Normal birth weight: belonging to the study area
* Low birth weight: being born at the national hospital

Exclusion Criteria:

* Overt illness
* Signs of vitamin A deficiency
* Previous BCG vaccination

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7600 (Actual)
Dates: Start 2004-11

PRIMARY OUTCOMES:
Mortality
Morbidity

SECONDARY OUTCOMES:
Adverse effects
Tuberculin reaction
BCG scarring
Growth
Vitamin A status
Cytokine responses
Malaria
Measles
Rotavirus
Respiratory syncytial virus (RSV) infection
All primary and secondary outcomes will be analysed for interactions between vitamin A and sex and last vaccine received.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Schaltz-Buchholzer F, Berendsen M, Roth A, Jensen KJ, Bjerregaard-Andersen M, Kjaer Sorensen M, Monteiro I, Aaby P, Stabell Benn C. BCG skin reactions by 2 months of age are associated with better survival in infancy: a prospective observational study from Guinea-Bissau. BMJ Glob Health. 2020 Sep;5(9):e002993. doi: 10.1136/bmjgh-2020-002993. PMID 32978212
- [Derived] Schaltz-Buchholzer F, Biering-Sorensen S, Lund N, Monteiro I, Umbasse P, Fisker AB, Andersen A, Rodrigues A, Aaby P, Benn CS. Early BCG Vaccination, Hospitalizations, and Hospital Deaths: Analysis of a Secondary Outcome in 3 Randomized Trials from Guinea-Bissau. J Infect Dis. 2019 Jan 29;219(4):624-632. doi: 10.1093/infdis/jiy544. PMID 30239767
- [Derived] Benn CS, Martins CL, Fisker AB, Diness BR, Garly ML, Balde I, Rodrigues A, Whittle H, Aaby P. Interaction between neonatal vitamin A supplementation and timing of measles vaccination: a retrospective analysis of three randomized trials from Guinea-Bissau. Vaccine. 2014 Sep 22;32(42):5468-74. doi: 10.1016/j.vaccine.2014.07.090. Epub 2014 Aug 13. PMID 25131735
- [Derived] Benn CS, Diness BR, Balde I, Rodrigues A, Lausch KR, Martins CL, Fisker AB, Aaby P. Two different doses of supplemental vitamin A did not affect mortality of normal-birth-weight neonates in Guinea-Bissau in a randomized controlled trial. J Nutr. 2014 Sep;144(9):1474-9. doi: 10.3945/jn.114.192674. Epub 2014 Jul 2. PMID 24991044
- [Derived] Biering-Sorensen S, Fisker AB, Ravn H, Camala L, Monteiro I, Aaby P, Benn CS. The effect of neonatal vitamin A supplementation on growth in the first year of life among low-birth-weight infants in Guinea-Bissau: two by two factorial randomised controlled trial. BMC Pediatr. 2013 May 23;13:87. doi: 10.1186/1471-2431-13-87. PMID 23702185
- [Derived] Benn CS, Fisker AB, Napirna BM, Roth A, Diness BR, Lausch KR, Ravn H, Yazdanbakhsh M, Rodrigues A, Whittle H, Aaby P. Vitamin A supplementation and BCG vaccination at birth in low birthweight neonates: two by two factorial randomised controlled trial. BMJ. 2010 Mar 9;340:c1101. doi: 10.1136/bmj.c1101. PMID 20215360